CLINICAL TRIAL: NCT02175394
Title: An Open, Two-period, Fixed-sequence, Phase I Trial to Evaluate the Effect of Multiple Doses of BI 1356 on the Multiple-dose Pharmacokinetics of a Combination of Ethinylestradiol and Levonorgestrel
Brief Title: Effect of Multiple BI 1356 Doses of on the Multiple-dose Pharmacokinetics of a Combination of Ethinylestradiol and Levonorgestrel in Healthy Female Premenopausal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1218.44
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination; Linagliptin

ARMS (2):
- Microgynon® (Active Comparator): Microgynon® once daily during period 1 (day 1 to day 14)
  Interventions: Drug: Microgynon®
- Microgynon® and BI 1356 (Experimental): Microgynon® combined with BI 1356, once daily during period 2 (day 15 to day 21)
  Interventions: Drug: Microgynon®; Drug: BI 1356

INTERVENTIONS:
Drug: Microgynon®
Drug: BI 1356
  Arms: Microgynon® and BI 1356

SUMMARY:
The objective was to investigate the effect of multiple oral doses of 5 mg BI 1356 on the steady-state pharmacokinetics of ethinylestradiol (EE) and levonorgestrel (LNG), the components of Microgynon®

ELIGIBILITY:
Inclusion Criteria:

* Healthy premenopausal female subjects as determined by the results of screening based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), heart rate (HR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Age 18 - 40 years
* BMI 18.5 - 27 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation
* Gynaecological examination without relevant findings

Exclusion Criteria:

* Any finding of the medical examination deviating from normal and of clinical relevance. Systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (greater than 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to day 1 or during the trial
* Use of antibiotics and drugs known to inhibit or induce cytochrome P450 enzymes, especially CYP3A4, within one month prior to study day 1 or during the trial (CYP3A4 inhibitors are for example azole antimycotics, macrolides, CYP3A inducers are for example St. John's Wort or certain anticonvulsants)
* Participation in another trial with an investigational drug within two months prior to day 1 or during the trial
* Regular smokers of more than two cigarettes daily
* Drug or alcohol abuse (more than 20 g alcohol/day)
* Blood donation (more than 100 mL within four weeks prior to day 1)
* Excessive physical activities within 48 hours prior to day 1)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* Positive pregnancy test, pregnancy or planning to become pregnant within 2 months of study completion, or lactation
* No use of an additional contraceptive method until 6 weeks after last study drug administration, i.e. barrier method, sexual abstinence, non-hormone-containing intrauterine device (IUD), surgical sterilisation (incl. hysterectomy) or vasectomized partner
* Use of oral contraceptive-containing intrauterine device, depot injection or contraceptive implants
* Existing or a history of confirmed venous thromboembolism (VTE), family history of idiopathic VTE and other known risk factors for VTE. Existing or previous arterial thrombotic or embolic processes, conditions which predispose to them e.g. disorders of the clotting processes, valvular heart disease and atrial fibrillation
* Relevant varicosis
* History of migraine
* History of liver disease, i.e. disturbances of liver function, jaundice or persistent itching during a previous pregnancy, Dubin-Johnson syndrome, Rotor syndrome, previous or existing liver tumours
* Clinically relevant cycle anomalies and dysmenorrhoea within the last 12 months
* Usual menstrual cycle duration outside of a 26-32 days range

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of ethinylestradiol and levonogestrel (Microgynon®) in plasma over the dosing interval at steady-state (AUCτ,ss) | On day 14 and on day 21
Maximum measured concentration of ethinylestradiol and levonogestrel (Microgynon®) in plasma at steady state (Cmax,ss) | On day 14 and on day 21

SECONDARY OUTCOMES:
Time from last dosing to the maximum measured concentration of EE and LNG in plasma at steady state (tmax,ss) | Up to day 22 after start of treatment
Apparent clearance of EE and LNG in plasma following extravascular administration at steady state (CL/F,ss) | Up to day 22 after start of treatment
Apparent volume of distribution of EE and LNG during the terminal phase λz at steady state following extravascular administration (Vz/F,ss) | Up to day 22 after start of treatment
Terminal half-life of EE and LNG in plasma at steady state (t1/2,ss) | Up to day 22 after start of treatment
Terminal rate constant of EE and LNG in plasma at steady state (λz,ss) | Up to day 22 after start of treatment
Mean residence time of EE and LNG in the body at steady state after oral administration (MRTpo,ss) | Up to day 22 after start of treatment
Pre-dose plasma concentrations of EE and LNG for attainment of steady state | Up to day 21 after start of Microgynon® treatment
Pre-dose plasma concentration of BI 1356 for attainment of steady state | Day 15 up to 7 days after start of BI 1356 treatment (day 21)
Plasma concentration of BI 1356 | Day 21
Number of patients with adverse events | Up to 14 weeks
Number of patients with clinically relevant changes in vital signs (BP, HR) | Up to 14 weeks
Number of patients with clinical relevant changes in laboratory evaluation (haematology, clinical chemistry and urinalysis) | Up to 14 weeks
Number of patients with clinically relevant changes in ECG recordings | Up to 14 weeks
Assessment of global tolerability by the investigator, a 4-point scale | Up to day 14 after last administration of study drug on day 21